CLINICAL TRIAL: NCT05766202
Title: The Development and Feasibility of Fear of Childbirth Intervention Aiming to Reduce Fear in Pregnant Multiparas: a Mixed Methods Study
Brief Title: The MOTIVE (Multiparas Overcoming Childbirth Fear Through Intervention and Empowerement) Feasibility Trial
Acronym: MOTIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University (Other)
Collaborators: Finnish Institute for Health and Welfare (Other Government); Metropolia University of Applied Sciences (Other); Kanta-Häme Central Hospital (Other Government)
Responsible Party: Principal Investigator, Laura Sandström, Principal Investigator, Tampere University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ETL-R22124H
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Fear of Childbirth; Anxiety; Depression
Keywords: Multipara; Psychoeducation; Prenatal class; Midwife; Psychiatric nurse
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pilot intervention for multiparas with fear of childbirth (Other): A group intervention with four meetings and one telephone call.
  Interventions: Other: An group intervention for multiparas with fear of childbirth

INTERVENTIONS:
Other: An group intervention for multiparas with fear of childbirth — The intervention consists of 4 group meetings, three during pregnancy and once after giving birth. It also includes a phone call.

SUMMARY:
The purpose of the study is to develop and pilot an intervention for the treatment of fear of childbirth for multiparas and to evaluate the feasibility of the intervention in the treatment of fear of childbirth in multiparas.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* understands finnish language
* has self reported fear of childbirth
* is a multipara
* under 35 weeks pregnant
* willingness to participate in the study

Exclusion Criteria:

* openly psychotic
* at risk of suicide
* serious substance abuse problems

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 19 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Change of Fear of Childbirth from baseline to pregnancy week 36 to 8 weeks after birth | Baseline, week 36 of pregnancy and 8 weeks after birth
  The FOBS (Fear of Birth scale) is a validated, self-reported instrument assessing fear of childbirth. Possible scores range from 0 (no fear) to 100 (worst possible fear). Change= (week 36 score - baseline score and 8 weeks after birth - baseline).

SECONDARY OUTCOMES:
Depression | Baseline, week 36 of pregnancy and 8 weeks after birth
  EPDS (Edinburgh postnatal depression scale) is a validated, self-reported instrument assessing depression.Change= (week 36 score - baseline score and 8 weeks after birth - baseline). Possible scores range from 0 to 30 points. A higher score pointing towards a worse outcome.
Anxiety | Baseline, week 36 of pregnancy and 8 weeks after birth
  HADS-A (Hospital Anxiety and depression scale - anxiety) is a validated, self-reported instrument assessing anxiety. Change= (week 36 score - baseline score and 8 weeks after birth - baseline).Possible scores range from 0 to 21 points. A higher score pointing towards a worse outcome.
Childbirth experience | Only one measurement point, at 8-weeks after birth.
  CPS (Childbirth perception scale) is a validated, self-reported instrument assessing childbirth experience. Possible scores range from 0 to 48 points. A higher score pointing towards a worse outcome.
Pregnancy related anxiety | Baseline and week 36 of pregnancy
  PRAQ-R2 (Pregnancy Related Anxiety Questionnaire for multiparas) is a validated, self-reported instrument assessing pregnancy related anxiety. Possible scores range from 10 to 50 points. A lower score pointing towards a worse outcome.
Maternal childbirth experience | Only one measurement point, at 8-weeks after birth.
  VAS (the visual analogue scale) is a ten-point horizontal line with verbal anchors at the extremes of the scale, where higher scores mean better outcomes. The minimum value is 1, and maximum value is 10. VAS has been used to measure the childbirth experience or satisfaction with the childbirth experience in various studies. In addition, VAS has been successfully tested against more detailed measurement instruments, such as the childbirth experience questionnaire (CEQ) and the Wijma Delivery Expectations / Experience Questionnaire (WDEQ-B).

CONTACTS AND LOCATIONS:
Overall Officials: Laura Sandström, MHSc, Principal Investigator — Tampere University
Locations (1):
- Kanta-Hämeen Keskussairaala, Hämeenlinna, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sandstrom L, Kaunonen M, Huhtala H, Aho AL. Evaluating a Group-Based Intervention Addressing Fear of Childbirth in Multiparous Pregnant Women: A Mixed Methods Feasibility Study. J Adv Nurs. 2025 May 23. doi: 10.1111/jan.17073. Online ahead of print. PMID 40405826